CLINICAL TRIAL: NCT03235986
Title: A Randomized, Open, Multinational, Multicentre,2-Part Study In Spontaneously Breathing Preterm Neonates With Mild To Moderate Respiratory Distress Syndrome (RDS) To Investigate The Safety, Tolerability And Efficacy Of Inhaled Nebulised Poractant Alfa (Porcine Surfactant, Curosurf®) In Comparison With Nasal Continuous Positive Airway Pressure (nCPAP) Alone
Brief Title: A Study To InvestigateThe Safety, Tolerability And Efficacy Of Nebulised Curosurf® In Preterm Neonates With Respiratory Distress Syndrome (RDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in the benefit-risk balance
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCD-01534CA1-01; 2016-004547-36 (EudraCT Number)
Record Dates: First submitted 2017-07-26; First posted 2017-08-01 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neonatal Respiratory Distress Syndrome
Keywords: RDS
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Continuous Positive Airway Pressure; Single Person

STUDY DESIGN:
Intervention Model Description: Part I is an ascending dose scheme of IMP versus nCPAP alone. Part II is a parallel group with 2 doses of IMP versus nCPAP alone. In part II, one additional dose may be administered between 3 and 12 hours after the start of the first dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nCPAP+ Nebulised Curosurf® (Experimental): Curosurf® administered through nebulization
  Interventions: Drug: nCPAP (nasal Continuous Positive Airway Pressure) + Nebulised Curosurf® (Part I); Drug: nCPAP (nasal Continuous Positive Airway Pressure) + Nebulised Curosurf® (Part II)
- nCPAP alone (control) (Other): Standard of care, respiratory support used also during experimental arms
  Interventions: Other: nCPAP (nasal Continuous Positive Airway Pressure) alone (Part I); Other: nCPAP (nasal Continuous Positive Airway Pressure) alone (Part II)

INTERVENTIONS:
Drug: nCPAP (nasal Continuous Positive Airway Pressure) + Nebulised Curosurf® (Part I) — Single ascending doses of Curosurf® administered through nebulisation to neonates receiving nCPAP (Part I)
  Arms: nCPAP+ Nebulised Curosurf®
Drug: nCPAP (nasal Continuous Positive Airway Pressure) + Nebulised Curosurf® (Part II) — Two doses of Curosurf® administered through nebulisation to neonates receiving nCPAP (Part II)
  Arms: nCPAP+ Nebulised Curosurf®
Other: nCPAP (nasal Continuous Positive Airway Pressure) alone (Part I) — Nasal continuous positive airway pressure alone
  Arms: nCPAP alone (control)
Other: nCPAP (nasal Continuous Positive Airway Pressure) alone (Part II) — nasal continuous positive airway pressure alone
  Arms: nCPAP alone (control)

SUMMARY:
The present study will mainly aim at investigating the safety, tolerability and efficacy of different escalating single doses administration of nebulised Curosurf®, in preterm neonates with RDS (Respiratory Distress Syndrome) during nCPAP.

DETAILED DESCRIPTION:
The study will be conducted in spontaneously breathing preterm neonates with mild to moderate RDS and will consist of two parts:

Part I, with the objective to assess the safety and tolerability of single ascending doses of nebulised Curosurf® ; Part II, with the objective to compare the efficacy of nebulised Curosurf®, administered at two selected doses from part I, during nCPAP, versus nCPAP alone in terms of incidence of respiratory failure in the first 72 hours of life.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained by parents/legal representative (according to local regulation) prior to or after birth
2. Inborn neonates from 28+0 to 32+6 weeks of gestational age (GA), spontaneously breathing and stabilised on nCPAP
3. Clinical course consistent with RDS.
4. Receiving CPAP pressure 5-8 centimeter of water (cm H2O) and fraction of inspired oxygen (FiO2) between 0.25 and 0.40 to maintain saturation of peripheral oxygen (SpO2) between 88% and 95% for at least 30 minutes. Randomization should occur between 60 minutes and 12 hours after birth.

Exclusion Criteria:

1. Early need for endotracheal intubation for cardiopulmonary resuscitation in delivery room or within 1 hour from birth because of severe RDS
2. Respiratory Distress not secondary to surfactant deficiency
3. Use of surfactant prior to study entry and need for endotracheal administration of any other treatment.
4. Major congenital anomalies.
5. Evidence of severe birth asphyxia
6. Mothers with prolonged rupture of the membranes
7. Presence of air leaks.
8. Presence of IVH (intraventricular hemorrhage ) ≥ III.
9. Hypotension or evidence of hemodynamic instability.
10. Any condition that, in the opinion of the Investigator, would place the neonate at undue risk.
11. Participation in another clinical trial

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Percentage of neonates with respiratory failure | in the first 72 hours of life
  Respiratory failure defined as: need for endotracheal surfactant administration and/or mechanical ventilation
Adverse Events | discharge or 36 weeks post menstrual age (PMA), whichever comes first
  Any untoward medical occurrence in a clinical trial neonate administered a medicinal product and which does not necessarily have a casual relationship with the treatment
Adverse Drug Reactions | discharge or 36 weeks post menstrual age (PMA), whichever comes first
  Any untoward and unintended responses to an investigational product related to any dose administered

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Dani, MD, Principal Investigator — Careggi Hospital, Florence (Italy)
Locations (1):
- Prof.Carlo Dani, Coordinating Investigator - Careggi Hospital, Florence (Italy), Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dani C, Talosi G, Piccinno A, Ginocchio VM, Balla G, Lavizzari A, Stranak Z, Gitto E, Martinelli S, Plavka R, Krolak-Olejnik B, Lista G, Spedicato F, Ciurlia G, Santoro D, Sweet D; CURONEB Study Group. A Randomized, Controlled Trial to Investigate the Efficacy of Nebulized Poractant Alfa in Premature Babies with Respiratory Distress Syndrome. J Pediatr. 2022 Jul;246:40-47.e5. doi: 10.1016/j.jpeds.2022.02.054. Epub 2022 Mar 5. PMID 35257740
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-004547-36/results